CLINICAL TRIAL: NCT06027619
Title: Short Contact Protocols to Reduce Pain During Treatment of Actinic Keratoses With 10% ALA Gel Red-light Photodynamic Therapy (PDT)
Brief Title: Short Contact Protocols to Reduce Pain During 10% ALA Gel Red-light Photodynamic Therapy of Actinic Keratoses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: The Cleveland Clinic (Other); Biofrontera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE4623
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-08

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratoses; Actinic Keratosis; Photodynamic Therapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Regimen A (Experimental): Apply topical aminolevulinic acid gel and incubate for 10 minutes prior to red light source
  Interventions: Drug: Topical aminolevulinate (10% ALA gel); Device: Red light illumination
- Regimen B (Experimental): Apply topical aminolevulinic acid gel and incubate for 20 minutes prior to red light source
  Interventions: Drug: Topical aminolevulinate (10% ALA gel); Device: Red light illumination
- Regimen C (Experimental): Apply topical aminolevulinic acid gel and incubate for 60 minutes prior to red light source
  Interventions: Drug: Topical aminolevulinate (10% ALA gel); Device: Red light illumination

INTERVENTIONS:
Drug: Topical aminolevulinate (10% ALA gel) — 10% ALA gel to the entire face, without occlusion, followed by a prespecified incubation period
  Other Names: Ameluz gel, 10% aminolevulinic acid
Device: Red light illumination — Illumination of red light of narrow spectrum of 635 nm with a light dose of approximately 37 J/cm2
  Other Names: BF-RhodoLED® Light Source

SUMMARY:
The goal of this clinical trial is to see if shorter Photodynamic Therapy (PDT) treatment times will still be effective at treating actinic keratoses (AK) while reducing or eliminating the pain that patients sometimes experience during conventional PDT treatment. The main questions it aims to answer are:

* Will the application of the nanoemulsion (10% ALA gel), in the absence of occlusion, still achieve significant inflammation and lesion clearance?
* Will shortened incubation times of Ameluz still achieve significant inflammation and lesion clearance?
* Will the new test regimens achieve reduced pain during illumination?
* Will the new test regimens be safe?

Participants will be randomly assigned to one of three treatment regimens, which will determine the length of time that the topical medication will incubate on the face before red light exposure in PDT treatments. The incubation period will be either 10 minutes, 20 minutes, or 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 10 actinic keratoses lesions on the face.
* Female subjects must not become pregnant during the study
* Subjects must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Pregnant or nursing.
* Using any topical treatment on their AKs; must stop at least one month prior.
* Currently undergoing treatment for other cancers with medical or radiation therapy.
* Patients with a known hypersensitivity to 5-aminolevulinic acid or any component of the study material.
* Patients with history of a photosensitivity disease, such as porphyria cutanea tarda.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward V Maytin, M.D. Ph.D., Principal Investigator — Cleveland Clinic, Dermatology and Plastic Surgery Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Dermatology and Plastic Surgery Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available 12/2024

REFERENCES:
- [Derived] Johnson JS, Hanna J, Nowacki AS, Anand S, Shen AS, Maytin EV. Painless PDT using 10% aminolevulinate gel and red light: A pilot clinical trial of short-contact protocols to reduce discomfort during illumination. Photodiagnosis Photodyn Ther. 2025 Aug;54:104698. doi: 10.1016/j.pdpdt.2025.104698. Epub 2025 Jun 26. PMID 40581198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 10 subjects are enrolled for each of the study arms A, B, and C.
Period: Overall Study
Arm/Group | Regimen A | Regimen B | Regimen C
Started | 10 | 10 | 10
Completed | 10 | 10 | 9
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A | Regimen B | Regimen C | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (7.4) | 69.9 (7.0) | 71.2 (5.8) | 70.1 (0.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 4
  Male | 9 | 10 | 7 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 9 | 9 | 27
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 10 | 10 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
History of skin cancer [Count of Participants; unit: Participants] | 9 | 8 | 7 | 24
AK lesions [Mean (Standard Deviation); unit: Lesions] | 54.8 (24.3) | 37.1 (17.3) | 46.3 (17.3) | 46.07 (8.85)
AKs previously [Count of Participants; unit: Participants] | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Treatment Efficacy Based on Participant AK Lesion Clearance
Description: To test the hypothesis that a short-contact PDT protocol with Ameluz and red light will produce lesion clearance outcomes that are statistically non-inferior to the traditional, painful protocol. This will be measured by Clinical Efficacy, which will be based on the AK lesion counts and lesion clearance rate after two treatments.
Time Frame: Lesion clearance at Visit 3 (month 2) and at Visit 4 (month 6)
Measure: Number; unit: percentage of AK lesions
Units Other Than Participants: Lesions
Arm/Group | Regimen A | Regimen B | Regimen C
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (Lesions) | 10 | 10 | 9
percentage of AK lesions
  Lesion clearance rate at Visit 3 | 59 | 34 | 43
  Lesion clearance rate at Visit 4 | 76 | 74 | 82

2. Primary Outcome: Differences in Pain Level Reported Throughout Exposure to Red Light
Description: Pain will be reported by the participants during illumination will be measured on a subjective 11-point visual-analog scale (VAS scale 0= no pain, 10 = intolerable pain)
Time Frame: Pain measured during illumination with red light (during a 10 min period) at Visit 1 (Day 3) and at Visit 3 (Month 2)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Regimen A | Regimen B | Regimen C
Number analyzed (Participants) | 10 | 10 | 9
score on a scale
  Pain at visit 1 | 0.70 (0.32) | 0.10 (0.11) | 4.7 (0.65)
  Pain at visit 3 | 0.20 (0.21) | 0.30 (0.16) | 2.22 (0.68)

3. Secondary Outcome: Patient Satisfaction Survey as Measured by Treatment Outcome Score
Description: Treatment score on a scale of 0 to 5, where 0 indicates extremely dissatisfied and 5 indicates extremely satisfied.
Time Frame: 6 months
Measure: Number; unit: percentage of patients
Arm/Group | Regimen A | Regimen B | Regimen C
Number analyzed (Participants) | 10 | 10 | 9
percentage of patients
  Percentages of patients giving a score of 5 | 80 | 60 | 89
  Percentages of patients giving a score of 4 | 10 | 30 | 11
  Percentages of patients giving a score of 3 | 10 | 10 | 0
  Percentages of patients giving a score of 2 | 0 | 0 | 0
  Percentages of patients giving a score of 1 | 0 | 0 | 0

4. Secondary Outcome: Patient Satisfaction Survey as Measured by Cosmetic Outcome Score
Description: Cosmetic score on a scale of 0 to 5, where 0 indicates extremely dissatisfied and 5 indicates extremely satisfied.
Time Frame: At month 6
Measure: Number; unit: percentage of patients
Arm/Group | Regimen A | Regimen B | Regimen C
Number analyzed (Participants) | 10 | 10 | 9
percentage of patients
  Percentage of participants giving a score of 5 | 70 | 50 | 89
  Percentage of participants giving a score of 4 | 20 | 40 | 0
  Percentage of participants giving a score of 3 | 10 | 10 | 11
  Percentage of participants giving a score of 2 | 0 | 0 | 0
  Percentage of participants giving a score of 1 | 0 | 0 | 0

5. Secondary Outcome: Number of Participant Reported Adverse Events and Side Effects
Description: Overall AE Profile and Safety of treatment will be measured using an Adverse Events- Patients' side effects log and Investigator assessment.
Time Frame: Up to 6 days (Day 6) after Visit 1
Measure: Number; unit: Number of events
Arm/Group | Regimen A | Regimen B | Regimen C
Number analyzed (Participants) | 9 | 10 | 9
Number of events
  Adverse events | 0 | 0 | 2
  Side effects | 9 | 10 | 9

ADVERSE EVENTS:
Time Frame: Serious adverse events that occur from signing of informed consent through 30 days after the last dose of treatment, up to 6 months
Arm/Group | Regimen A | Regimen B | Regimen C
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (N=10) | Regimen B (N=10) | Regimen C (N=10)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT06027619/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT06027619/ICF_001.pdf